CLINICAL TRIAL: NCT05524610
Title: Stakeholder-Engaged Development and Evaluation of a Screening Approach for Sexual Dysfunction in Adolescent and Young Adult Patients With and Surviving Childhood Cancer
Brief Title: Development and Evaluation of a Screening Approach for Sexual Dysfunction in AYA Patients With and Surviving Childhood Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-0709.ccc; K08CA263192 (NIH)
Record Dates: First submitted 2022-08-25; First posted 2022-09-01 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Pediatric Cancer; Survivorship
Keywords: Cancer Survivor; Cancer Patient; Young Adult
MeSH Terms: conditions — Neoplasms | interventions — National Institutes of Health (U.S.)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Implementation of Routine Sexual Function Screening (Baseline) (No Intervention): This arm will include patients with and surviving cancer who are seen during the Pre-Implementation study period. It will include patients diagnosed prior to age 18 years and 15-24 years old at the time of study. Patients will be approached by research personnel at the end of each visit for participation in a survey. The pre-implementation survey will assess sexual function communication and patient satisfaction. In addition, medical record data abstraction of clinical care related to sexual health and function will be collected.
- Post-Implementation of Routine Sexual Function Screening (Experimental): This arm will include patients with and surviving cancer who are seen during the Post-Implementation study period, once the routine sexual function screening intervention has been implemented. It will include patients diagnosed prior to age 18 years and 15-24 years old at the time of study. Patients will be approached by research personnel at the end of each visit for participation in a survey. The post-implementation survey will assess sexual function communication and patient satisfaction, as well as measures of acceptability, feasibility, and appropriateness of the intervention. In addition, medical record data abstraction of clinical care related to sexual health and function will be collected.
  Interventions: Behavioral: Sexual Function Screening Approach

INTERVENTIONS:
Behavioral: Sexual Function Screening Approach — The screening approach will consist of:
  1. Standardized use of the PROMIS SexFS Brief in a clinic setting. This tool assesses sexual interest/desire, arousal, discomfort/pain, climax, and satisfaction, among other SD concerns and has comparable sex-specific versions. It has been validated in adult cancer populations.
  2. An implementation package to aid in successful implementation. The implementation package will be finalized in the non-trial portion of this study, which will include iterative intervention adaptation. The protocol will be amended as needed to include any relevant updates to the screening approach. Some components may vary per site.
  Other Names: National Institute of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS®) Sexual Function and Satisfaction (SexFS) Brief v2.0 tool
  Arms: Post-Implementation of Routine Sexual Function Screening

SUMMARY:
Prior research determined adolescent and young adult-aged childhood cancer survivor (AYA-CCS) and medical provider acceptability of the SexFS Brief in a controlled research setting. Development of an acceptable, effective, and feasible screening approach will result in improved recognition of SD in AYA patients with and surviving childhood cancer.

DETAILED DESCRIPTION:
Detailed Description:

To adhere to National Comprehensive Cancer Network (NCCN) Adolescent and young adult (AYA) and Survivorship Guidelines, the Investigator will be developing and implementing a standardized screening approach for sexual function using the Patient Reported Outcome Measurement Information System (PROMIS) for Sexual Function and Satisfaction (SexFS) Brief. The overarching goal of this proposal is to develop and pilot test a patient-centered approach to assessing AYA patients with and surviving childhood cancer (age 15-24) for SD.

Prior to the clinical trial, Aim 1 of this study will integrate patient and provider feedback to refine an approach to standardized sexual function screening. Once Aim 1 has been completed, the study protocol will be amended to update intervention details prior to proceeding with implementation across all clinics as routine clinical care.

Aims 2 and 3 involve a pilot type 1 hybrid effectiveness-implementation trial using a pre-post design. Prior to implementation of the intervention, data on sexual function screening and patient satisfaction will be collected through surveys and medical record review. Subsequently, the sexual function screening intervention will be implemented clinic-wide as standard of care for patients age 15-24 years with or surviving childhood cancer. Following implementation of the screening approach, post-implementation data (effectiveness and implementation outcomes) will be collecting via survey and EHR review in consenting patients. After effectiveness data collection is complete, implementation outcomes will also be assessed via surveys and interviews with consenting provider stakeholders.

ELIGIBILITY:
Inclusion Criteria

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be aged 15-24 years old at the time of enrollment
4. Patients with or surviving of cancer (must be found in the International Classification of Diseases for Oncology (ICD-O) and have a behavior code ≥2)
5. Must have received cancer-directed therapy with at least one of the following:

   * Chemotherapy: any anticancer drug to treat the cancer diagnosis including immunotherapy
   * Radiotherapy: any radiotherapy to treat the cancer diagnosis
   * Surgery: any surgery to remove cancer including partial or total resections. Biopsies are not considered surgery.
6. Cancer must have been diagnosed before the age of 18 years
7. Patient must have an appointment at one of four clinical sites: CHCO HOPE Survivorship Program, CHCO Oncology Clinic, CHCO Neuro-Oncology Clinic, Seattle Children's Hospital Survivorship Program

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Unable to read and speak English
2. Patients who did not receive cancer-directed therapy
3. Insufficient cognitive functioning to complete study measures, as determined by patient's
4. Participation in intervention development
5. Patient is at end of life or on hospice, as determined by primary oncologist
6. Patients who did not undergo sexual function screening within 1 month of being due will be excluded from implementation outcomes measurement
7. Patient is at end of life or on hospice, as determined by primary oncologist

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 205 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of sexual function communication before and after intervention implementation | 5 years
  Comparison of pre- and post- intervention percentage of patients reporting that his/her provider has communicated with them about sexual function Subjects will report (yes or no) via survey after their healthcare visit.

SECONDARY OUTCOMES:
Comparison of patient satisfaction before and after intervention implementation | 5 years
  Comparison of pre- and post-intervention rating of patient satisfaction with sexual function communication. Subjects will report via survey after their healthcare visit. This will be rated on a 10-point scale with 10 being very satisfied and 0 being not at all satisfied.
Comparison of healthcare needs being met before and after intervention implementation | 5 years
  Comparison of pre- and post-intervention percentage of patients with self-identified sexual function needs reporting that this need was met. Subjects will report (yes or no) via survey after their healthcare visit. .
Reach - proportion of eligible patients who completed sexual function screening | 5 years
  Record abstraction evaluating the proportion of eligible patients who completed sexual function screening
Representativeness - sociodemographic characteristics of patients who received and did not receive screening | 5 years
  Comparison of sociodemographic characteristics between eligible patients who did versus did not receive sexual function screening.
Adoption of the screening tool by medical stakeholders (self-reported results review) | 5 years
  Medical stakeholder survey score of a 5-point scale (1=never, 5=every time) on a survey at the conclusion of the study, asking how often they reviewed sexual function screening results with relevant patients
Adoption of the screening tool by medical stakeholders (self-reported results discussion) | 5 years
  Medical stakeholder survey score of a 5-point scale (1=never, 5=every time) on a survey at the conclusion of the study, asking how often they discussed results with patients
Patient-reported acceptability of the sexual function screening approach | 5 years
  Patients will complete a study-specific acceptability survey consisting of several questions on a 5-point scale (0=low acceptability, 5=high acceptability)
Provider-reported acceptability of the sexual function screening approach | 5 years
  Providers will complete the Acceptability of Intervention Measure (AIM), adapted for this study, which consists of several questions on a 5-point scale (0=low acceptability, 5=high acceptability)
Patient-reported appropriateness of the sexual function screening approach | 5 years
  Patients will complete a study-specific appropriateness survey consisting of several questions on a 5-point scale (0=low acceptability, 5=high acceptability)
Provider-reported appropriateness of the sexual function screening approach | 5 years
  Providers will complete the Intervention Appropriateness Measure (IAM), adapted for this study, which consists of several questions on a 5-point scale (0=low appropriateness, 5=high appropriateness)
Patient-reported feasibility of the sexual function screening approach | 5 years
  Patients will complete a study-specific feasibility survey consisting of several questions on a 5-point scale (0=low feasibility, 5=high feasibility)
Provider-reported feasibility of the sexual function screening approach | 5 years
  Providers will complete the Feasibility of Intervention Measure (FIM), adapted for this study, which consists of several questions on a 5-point scale (0=low feasibility, 5=high feasibility)
Evaluate implementation of the standardized screening approach by fidelity (patient-reported) | 5 years
  Patients will respond regarding whether or not they experienced key components (Fidelity Checklist) of the intervention.
Evaluate implementation of the standardized screening approach by fidelity (direct observation) | 5 years
  The study team will evaluate whether key components of the intervention (Fidelity Checklist) are completed via direct observation in 10% of patients across sites.
Contextual factors influencing implementation success | 5 years
  Qualitative description of themes, barriers and facilitators to implementation will be determined via interviews with medical providers after completion of patient enrollment.

OTHER OUTCOMES:
Referral patterns for sexual function concerns | 5 years
  Comparison the referral patterns before and after implementation of the sexual function screening approach (exploratory)
Incidence of documented sexual function concerns | 5 years
  Comparison the documentation about sexual function concerns before and after implementation of the sexual function screening approach (exploratory)
Adoption, as measured by proportion of results that are viewed (objective measure) | 5 years
  Proportion of answered sexual function screening surveys that show evidence of having been viewed (i.e. electronic health record (EHR) clicks)
Reach - Reason for missed screening | 5 years
  For patients who do not receive screening within 1 month of it being due, reach will be explored via a single multiple choice question to the medical team inquiring into the reasoning for missed screening
Adaptations to the sexual function screening approach | 5 years
  Qualitative description of documented adaptations to the screening approach as they occur throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Demedis, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Childrens Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No